CLINICAL TRIAL: NCT04055129
Title: 17b-Estradiol Induced Effects on Anterior Cruciate Ligament Laxity, Lower Extremity Biomechanics and Neuromuscular Activation Patterns in Females During Landing Activities
Brief Title: Hormone Induced Effects on Ligament Laxity and Lower Extremity Motor Control
Status: Completed | Type: Observational
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Principal Investigator, Kayla Smith PT, MSPT, DSc, University of St. Augustine for Health Sciences, University of St. Augustine for Health Sciences
Other Study IDs: 0430-018
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hormone Influence on Ligament Laxity and Motor Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva samples to be frozen and sent to lab for amount of estrogen analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Birth Control: Hormone levels controlled with subject on birth control pill
  Interventions: Other: No interventions
- Non-Birth Control: Hormone (estrogen) levels not controlled but monitored for levels of estrogen at two points in menstrual cycle (Follicular and ovulatory phases)
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — Observational. Data will be gathered and analyzed on ligament laxity, EMG, kinetics and kinematics during a landing and jumping activity

SUMMARY:
The purpose of this study is to expand on previous knowledge of the hormonal effects, specifically estrogen, on ligament laxity, motor control and timing of muscle activation in females. A significant amount of research has previously been done on the effects of estrogen throughout the menstrual cycle on ligament laxity with some showing a correlation of increased estrogen levels with increased ligament laxity. There have also been several studies that investigated muscle activation and ground reaction forces as related to hormone levels and stages of the menstrual cycle. A recent systematic review found a lack of research investigating muscle activation timing as related to hormonal changes despite theories suggesting muscle function including timing could be an explanation as to the potential causes for increased ACL injury correlated with the luteal phase of the menstrual cycle. The aim of this study is therefore to investigate whether hormonal changes throughout the menstrual cycle correlate with changes in ligament laxity, motor control, muscle activation and timing.

This study will be a longitudinal controlled study with two groups both containing females ages 18-35 years of age. The subjects will be placed into either the Experimental Group (no birth control) or the Control Group (on birth control) depending on the status of their contraceptive use.

DETAILED DESCRIPTION:
The purpose of this study is to expand on previous knowledge of the hormonal effects, specifically estrogen, on ligament laxity, motor control and timing of muscle activation in females. A significant amount of research has previously been done on the effects of estrogen throughout the menstrual cycle on ligament laxity with some showing a correlation of increased estrogen levels with increased ligament laxity. There have also been several studies that investigated muscle activation and ground reaction forces as related to hormone levels and stages of the menstrual cycle. A recent systematic review found a lack of research investigating muscle activation timing as related to hormonal changes despite theories suggesting muscle function including timing could be an explanation as to the potential causes for increased ACL injury correlated with the luteal phase of the menstrual cycle. The aim of this study is therefore to investigate whether hormonal changes throughout the menstrual cycle correlate with changes in ligament laxity, motor control, muscle activation and timing.

This study will be a longitudinal controlled study with two groups both containing females ages 18-35 years of age. The subjects will be placed into either the Experimental Group (no birth control) or the Control Group (on birth control) depending on the status of their contraceptive use. To ensure subject privacy, all investigators will be blinded to which group the subject is in during data collection except for the primary investigator who will do the initial meeting with the subjects to go through the informed consent, determine phase of menstrual cycle, and allocate the subject to a group based on their contraceptive use. From this point on, the subject will be identified by a subject number and all data intake and analysis will be done with the number identifier. Ovulation cycle will be identified by a self-administered ovulation kit, hormonal samples of Estrogen will be obtained by a saliva sample and sent to Salimetrics lab for analysis. Dependent measures will include recording subject single and double-leg jump off a 12- inch block and landing on a force plate to record muscle timing and ground reaction forces upon landing. Electromyography will be used to measure muscle activation timing of the quadriceps, hamstrings, gluteus maximus, gluteal medius, and gastrocnemius muscles. A 3-D measuring system will record trunk and hip flexion, femoral internal rotation angle, and knee flexion, extension and valgus angles. Finally, ligament laxity will be measured with a knee arthrometer (KT1000 or similar) device to record tibial anterior translation. Each subject will be tested, and each variable above will be recorded 2 separate times corresponding to 2 main phases in the menstrual cycle (Follicular and Ovulatory phases).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-35 years of age
* Group A) Not on Oral Contraceptive Group (NOC):

  * Regular menstrual cycle for a minimum of 2 consecutive months
  * No oral contraceptive birth control for a minimum of 6 months.
* Group B) Oral Contraceptive Group (OC):

  * Currently on oral hormone-based contraceptive intended to cease ovulation)

Exclusion Criteria:

* Previous lower extremity or spine injury
* Complaint of knee pain within past 6 months
* Irregular menstrual cycle (not consistently following a 28-32 cycle for a minimum of 2 months)
* Unable to meet physical demands of testing criterion:

  * Forward jump off 12- inch height step both legs and then single leg
  * Assume single leg-stance
  * Adhesive/electrode allergy
  * Pain or report of discomfort with any testing
  * Unable to produce saliva sample
  * Taking hormone replacements or medications known to cross-react with saliva sample and potentially give false data results (Fulvestrant/ Faslodex)
* History of pregnancy
* Smoker
* BMI >25
* Thyroid issues
* Connective tissue diseases (such as Ehlers-Danlos Syndrome, Marfan's Disease, Rheumatoid Arthritis)
* Excessive laxity of ACL (greater than 3 mm side to side anterior laxity measure on knee arthrometer)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 26 females on birth control, 26 not on birth control
Study Population: 52 healthy females (26 on birth control, 26 not on birth control), with healthy knees aged 18-35 years old.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Muscle activity for the following muscles: Quadriceps (vastus medialis and vastus lateralis), Hamstrings (semitendinosus, biceps femoris), gluteus maximus, gluteus medius, lateral gastrocnemius | July 01, 2021
  EMG recording to detect initiation of muscle activation for these muscles will be measured with EMG electrodes and software to detect when these muscles turn on and when they peak in their activity during a step down and jump activity.
Ground Reaction Force | July 01, 2021
  A force plate and computer program will be used to detect the ground reaction forces during a step down and jump activity

SECONDARY OUTCOMES:
Knee valgus, femoral internal rotation angle, knee flexion and extension angles | July 01,2019
  Lower extremity kinematics will be measured by using reflective markers and Simi 3D Motion capture system and markers to detect joint angle changes during a step down and jump activity (via computer software)
Laxity of ACL/ anterior tibial excursion | July 01, 2019
  Anterior displacement of tibia on femur will be measured using the GNRB devive which measures anteior displacement in millimeters with a computer generated force (Newtons) and reading (MM)

CONTACTS AND LOCATIONS:
Overall Officials: Kayla M Smith, Dsc, Principal Investigator — University of St. Augustine for Health Sciences
Locations (1):
- University of St. Augustine for Health Sciences, San Marcos, California, United States

IPD SHARING:
Plan to Share IPD: No